CLINICAL TRIAL: NCT06063811
Title: Characterization of Ventricular Tachycardia Ablation in End-stage Heart Failure Patients With Left Ventricular Assist Device
Brief Title: Ventricular Tachycardia Ablation in LVAD Patients
Acronym: CHANNELED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: CHANNELED-Registry
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Ventricular Tachycardia; End-stage Heart Failure; Ventricular Arrythmia; LVAD (Left Ventricular Assist Device)
Keywords: Catheter Ablation; VT Ablation in LVAD patients
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LVAD patients: Patients with end-stage heart failure with an LVAD implanted undergoing VT ablation.
  Interventions: Other: Ablation

INTERVENTIONS:
Other: Ablation — VT ablation

SUMMARY:
The CHANNELED-Registry is a multicenter retrospective study to (1) systematically assess the mechanism and origin of ventricular tachycardia in patients with end-stage heart failure carrying an left ventricular assist device (LVAD) and (2) to evaluate procedural parameters and outcome of ventricular tachycardia ablation in this special subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with end-stage heart failure with an LVAD implanted undergoing VT ablation

Exclusion Criteria:

* Patients <18 years, pregnant women, patients undergoing VT ablation without an LVAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with end-stage heart failure and an implanted LVAD which underwent ablation of ventricular tachycardia will be included in this retrospective observational study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Mechanism of ventricular tachycardia in LVAD patients (descriptive name of scale) | 12 month
  Assessment of the mechanism of VT in LVAD patients (e.g LVAD cannula related vs. related to substrate of underlying heart disease)
Number of patients with ventricular tachycardia recurrence in device interrogation (physiological parameter) | 12 month
  Assessment of VT recurrence after ablation: Device interrogation and readout of ICD Holter
Mortality (physiological parameter) | 12 month
  Assessment of mortality after VT ablation.
Heart failure Hospitalization (physiological parameter) | 12 month
  Assessment of Hospitalization for worsening of Heart Failure after VT ablation.

SECONDARY OUTCOMES:
Procedure duration (From groin puncture to sheath removal in minutes) | 12 month
  Evaluation of the duration of VT ablation procedures in LVAD patients
Fluoroscopy time (minutes) | 12 month
  Evaluation of the fluroscopy use (in minutes)
Radiofrequency energy used for ablation (in watts; e.g. 40 Watts) | 12 month
  Evaluation of the maximum RF-energy used for ablation
Number of patients suffering from intraprocedural complication (physiological parameter, e.g. hematoma) | 12 month
  Evaluation of intraprocedural complications of VT ablation

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lüker, MD, Principal Investigator — Heart Center University of Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Bruck JH, Hohendanner F, Heil E, Albert K, Duncker D, Estner H, Deneke T, Parwani A, Potapov E, Seuthe K, Wormann J, Sultan A, Schipper JH, Eckardt L, Doldi F, Lugenbiel P, Servatius H, Thalmann G, Reichlin T, Khalaph M, Guckel D, Sommer P, Steven D, Luker J. Characterization of ventricular tachycardia ablation in end-stage heart failure patients with left ventricular assist device (CHANNELED registry). Europace. 2025 Mar 28;27(4):euaf054. doi: 10.1093/europace/euaf054. PMID 40101155